CLINICAL TRIAL: NCT03439085
Title: A Phase 2, Open-Label Study to Evaluate Efficacy of Combination Treatment With MEDI0457 (INO-3112) and Durvalumab (MEDI4736) in Patients With Recurrent/Metastatic Human Papilloma Virus Associated Cancers
Brief Title: DNA Plasmid-encoding Interleukin-12/HPV DNA Plasmids Therapeutic Vaccine INO-3112 and Durvalumab in Treating Patients With Recurrent or Metastatic Human Papillomavirus Associated Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Project delays
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-0302; NCI-2018-00914 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2017-0302 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2018-02-14; First posted 2018-02-20 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-05

CONDITIONS: Human Papillomavirus-16 Positive; Human Papillomavirus-18 Positive; Metastatic Malignant Neoplasm; Recurrent Anal Canal Carcinoma; Recurrent Cervical Carcinoma; Recurrent Malignant Neoplasm; Recurrent Penile Carcinoma; Recurrent Vaginal Carcinoma; Recurrent Vulvar Carcinoma; Refractory Malignant Neoplasm; Stage IV Anal Cancer AJCC v8; Stage IV Cervical Cancer AJCC v8; Stage IV Penile Cancer AJCC v8; Stage IV Vaginal Cancer AJCC v8; Stage IV Vulvar Cancer AJCC v8; Stage IVA Cervical Cancer AJCC v8; Stage IVA Vaginal Cancer AJCC v8; Stage IVA Vulvar Cancer AJCC v8; Stage IVB Cervical Cancer AJCC v8; Stage IVB Vaginal Cancer AJCC v8; Stage IVB Vulvar Cancer AJCC v8
MeSH Terms: conditions — Neoplasm Metastasis; Anal Canal Carcinoma; Uterine Cervical Neoplasms; Recurrence; Penile Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Neoplasms; Anus Neoplasms | interventions — MEDI0457; VGX-3100; rocakinogene sifuplasmid; durvalumab; Immunoglobulin G; Disulfides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (INO-3112, durvalumab) (Experimental): Patients receive DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 IM and via electroporation at 1, 3, 7, and 12 weeks and durvalumab IV at 4, 8, and 12 weeks. Starting week 12, cycles repeat every 8 weeks for DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 and every 4 weeks for up to 13 doses of durvalumab in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: DNA Plasmid-encoding Interleukin-12/HPV DNA Plasmids Therapeutic Vaccine MEDI0457; Biological: Durvalumab

INTERVENTIONS:
Biological: DNA Plasmid-encoding Interleukin-12/HPV DNA Plasmids Therapeutic Vaccine MEDI0457 — Given IM and via electroporation
  Other Names: INO 3112; INO-3112; INO-3112 Vaccine; MEDI 0457; MEDI-0457; MEDI0457; VGX-3100 Plus INO-9012
Biological: Durvalumab — Given IV
  Other Names: Imfinzi; Immunoglobulin G1, Anti-(Human Protein B7-H1) (Human Monoclonal MEDI4736 Heavy Chain), Disulfide with Human Monoclonal MEDI4736 Kappa-chain, Dimer; MEDI-4736; MEDI4736

SUMMARY:
This phase II trial studies how well deoxyribonucleic acid (DNA) plasmid-encoding interleukin-12/human papillomavirus (HPV) DNA plasmids therapeutic vaccine INO-3112 and durvalumab work in treating patients with human papillomavirus associated cancers that have come back or spread to other places in the body. Vaccines made from a gene-modified virus may help the body build an effective immune response to kill tumor cells. Immunotherapy with monoclonal antibodies, such as durvalumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Giving DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 and durvalumab may work better in treating patients with human papillomavirus associated cancers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the anti-tumor activity of DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 (MEDI0457) in combination with durvalumab.

SECONDARY OBJECTIVES:

I. To determine the safety profile of MEDI0457 in combination with durvalumab in patients with recurrent/metastatic human papilloma virus (HPV) 16- or 18- associated cancer.

II. To evaluate the progression-free survival (PFS) and overall survival (OS) of patients with recurrent/metastatic incurable HPV-16/18 positive solid malignancies receiving the combination of MEDI0457and durvalumab.

III. To evaluate objective response rate (ORR) by immune-related criteria of the combination of MEDI0457 and durvalumab in patients with recurrent/metastatic incurable HPV-16/18 positive solid malignancies.

IV. To evaluate the disease control rate at 24 weeks.

EXPLORATORY OBJECTIVES:

I. To determine the cellular and humoral immune response to immunotherapy with MEDI0457 in combination with durvalumab,

II. To examine the correlation between anti tumor activity and biomarkers including:

IIa. HPV-specific cellular and humoral responses. IIb. Programmed death ligand 1 status. IIc. The number of tumor infiltrating lymphocytes, HPV 16/18 E6/E7 deoxyribonucleic acid (DNA) levels and HPV 16/18 E6/E7 DNA sequence in biopsy tissue and plasma.

III. To evaluate the pharmacokinetics and anti-drug antibodies (ADA) for durvalumab.

OUTLINE:

Patients receive DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 intramuscularly (IM) and via electroporation at 1, 3, 7, and 12 weeks and durvalumab intravenously (IV) at 4, 8, and 12 weeks. Starting week 12, cycles repeat every 8 weeks for DNA plasmid-encoding interleukin-12/HPV DNA plasmids therapeutic vaccine INO-3112 and every 4 weeks for up to 13 doses of durvalumab in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 90 days, every 3 months for 12 months, and then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with institutional guidelines.
* Are able and willing to comply with all study procedures.
* For patients who are not human immunodeficiency virus (HIV) positive, cervical, anal, penile, vulvar, or vaginal cancer positive for HPV-16 and/or HPV-18 by the institutionally approved assay. For patients who are HIV positive, histologically or cytologically confirmed diagnosis of cancer at any site that is positive for HPV-16 and/or HPV-18 by the institutionally approved assay. Tumors may be positive for more than 1 HPV subtype as long as HPV-16 and/or HPV-18 is present. Note: For the first 3 patients, only cervical, vulvar, or vaginal cancers will be enrolled.
* Patients with cancer that is refractory to standard therapy, that have either relapsed after standard therapy or has no standard therapy that increases survival by at least three months, and/or that are not curable by salvage approaches including resection and/or re-irradiation
* Has measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) with a minimum size of 10 mm by computed tomography (CT) scan, except lymph nodes which must have minimum short axis size of 15 mm (CT scan slice thickness no greater than 5 mm in both cases). Indicator lesions must not have been previously treated with surgery, radiation therapy, or radiofrequency ablation unless there is documented Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 progression in the lesion after such therapy.
* All patients must consent to pre-treatment biopsy of the tumor if it can be done safely (as judged by the investigator) during screening. Week 10 on-treatment biopsies will be required for a minimum 10 patients. After 10 paired biopsies have been obtained then week 10 on-treatment biopsy will be made optional.
* World Health Organization (WHO)/Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Hemoglobin >= 9 g/dL (Note: Note: No Transfusion within 7 days of beginning study treatment. Ongoing growth factor support is acceptable if on a stable dose for the past 56 days), within 28 days of day 0.

  * Cannot be met with recent blood transfusions or require ongoing growth factor support
* Absolute neutrophil count >= 1,000/mm^3, within 28 days of day 0.

  * Cannot be met with recent blood transfusions or require ongoing growth factor support
* Platelet count >= 100,000/mm^3 and no transfusion in prior 4 weeks, within 28 days of day 0.

  * Cannot be met with recent blood transfusions or require ongoing growth factor support
* Total bilirubin (TBL) =< 1.5 x upper limit of normal (ULN) except patients with documented Gilbert's syndrome (> 3 x ULN), within 28 days of day 0.
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 x ULN, within 28 days of day 0.
* Serum creatinine =< 2.0 mg/dL or creatinine clearance >= 40 mL/min (measured or calculated according to the method of Cockcroft and Gault), within 28 days of day 0.
* For human immunodeficiency virus (HIV)+ patients: documented HIV-1 infection with CD4 count > 200 cells/mm^3 and viral load < 75 copies/mL, within 28 days of day 0.

Exclusion Criteria:

* Any concurrent chemotherapy, investigational product (IP), biologic, or hormonal therapy for cancer treatment; receipt of any investigational or approved anticancer therapy (chemotherapy, targeted therapy, biologic therapy, monoclonal antibodies, etc.) within 21 days or 5 half lives, whichever is shorter, prior to the first dose of MEDI0457; concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Major surgical procedure or significant traumatic injury within 28 days before the first dose of study drug or anticipation of the need for major surgery during the course of study treatment.
* Any unresolved toxicity (National Cancer Institute Common Terminology Criteria for Adverse Event [CTCAE] version 4.03 [v4.03]) grade 2 or greater from previous anticancer therapy with the exception of alopecia, and the laboratory values defined in the inclusion criterion 8. Hearing loss of grade 3 or lower and peripheral neuropathy of grade 2 or lower is allowed. Subjects with grade >= 2 neuropathy will be evaluated on a case-by-case basis after consultation with the study physician. Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the study physician.
* Current or prior use of immunosuppressive medication within 14 days prior to first study dose, with the exception of intranasal and inhaled corticosteroids or systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or equivalent. Steroids as premedication for hypersensitivity reactions due to radiographic contrast agents are allowed.
* Patients requiring therapeutic anticoagulation and irreversible platelet inhibitors (e.g. clopidogrel, prasugrel, or ticagrelor). Low dose aspirin for cardiac prophylaxis is allowed.
* History of primary immunodeficiency.
* Patients who have had prior exposure to immune-mediated therapy, including but not limited to prior exposure to T-cell and natural killer cell directed therapy, anti-PD-1, anti-PD-L1, anti-CD137, and anti-CTLA4.
* History of allogeneic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g. colitis, ulcerative colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc.]). The following are exceptions to this criterion: patients with vitiligo or alopecia, patients with hypothyroidism (e.g. following Hashimoto syndrome) stable on hormone replacement, any chronic skin condition that does not require systemic therapy, patients without active disease in the last 5 years may be included but only after consultation with the study physician, and patients with celiac disease controlled by diet alone.
* Uncontrolled intercurrent illness, including, but not limited to, ongoing or active infection, uncontrolled hypertension, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events, or compromise the ability of the patient to give written informed consent.
* Patients with spinal cord compression or a history of leptomeningeal carcinomatosis. At the time of day 1 of the study, patients with central nervous system metastases must have been treated and must be asymptomatic and meet the following criteria. 1. No concurrent treatment, inclusive of, but not limited to, surgery, radiation, and/or corticosteroids. (Note: patients are allowed on systemic steroids unless these are being administered to manage central nervous system metastases); 2. Neurologic stability (lack of signs or symptoms greater than baseline prior to radiotherapy) until the time of dosing of MEDI0457; 3. For radiation treatment, patients must be: at least 14 days between last day of stereotactic radiosurgery or gamma-knife treatment and day 1 of protocol treatment, at least 28 days between last day of whole brain radiation therapy and day 1 of protocol treatment, and/or at least 14 days since last dose of corticosteroids and day 1 of protocol treatment.
* Patients with cardiovascular (CV) disease conditions including New York Heart Association class 3 or 4 congestive heart failure, unstable angina pectoris, or clinically important cardiac arrhythmias OR a recent (< 3 months) CV event, including myocardial infarction, unstable angina pectoris, or stroke.
* Mean QT interval corrected for heart rate (QTc) >= 470 ms calculated from electrocardiogram (ECG) using Fridericia's correction by manual read.
* Active tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and tuberculosis testing in line with local practice) infection.
* Presence of acute or chronic hepatitis B (hepatitis B virus [HBV]) or active hepatitis C (hepatitis C virus [HCV]). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBV surface antigen [HBsAg]) are eligible. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV ribonucleic acid (RNA).
* Receipt of live, attenuated vaccine within 30 days prior to study entry or the first dose of MEDI0457.

  * Note: patients, if enrolled, should not receive live vaccine during the study and up to 30 days after the last dose of IP.
* Other untreated coexisting HIV related malignancies.
* History of another primary malignancy except for: malignancy treated with curative intent and with no known active disease >= 2 years before the first dose of IP and of low potential risk for recurrence, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, or adequately treated carcinoma in situ without evidence of disease.
* Pregnant or breastfeeding female patients.
* Known allergy or hypersensitivity to study treatment or any of the study drugs excipients.
* Any medical condition that, in the opinion of the investigator, would interfere with evaluation of the study treatment or interpretation of patient safety or study results.
* Patients with active or prior digestive tract bleeding.
* Patients with uncontrolled seizures.
* Fewer than two acceptable sites exist for intramuscular (IM) injection and electroporation (EP) between the deltoid and lateral quadriceps muscles. Note: a site for injection/EP is not acceptable if there are tattoos or scars within 2 cm of the proposed injection/EP site or if there is implanted metal within the same limb. Any device implanted in the chest (e.g. cardiac pacemaker or defibrillator) excludes the use of the deltoid muscle on the same side of the body.
* Patients who are unable to provide informed consent, are incarcerated, or are unable to follow protocol requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2022-09-20 (Actual); Study Completion 2022-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael M Frumovitz, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on 11/14/2018 and closed to new patient entry on 08/12/2021. The study was terminated on 09/20/2022 and all recruitment was done in a medical clinic setting.
Groups:
- Treatment Group: Patients received 7 mg of MEDI0457 intramuscularly (weeks 1, 3, 7, 12, and every 8 weeks thereafter) and durvalumab 1500 mg intravenously every 4 weeks starting at week 4.
Period: Overall Study
Arm/Group | Treatment Group
Started | 41
Completed | 19
Not Completed | 22
Not completed — Death | 2
Not completed — Screen Failure | 20

BASELINE CHARACTERISTICS:
Arm/Group | Treatment Group
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 37
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 49 [28 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 30
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: Will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Will be estimated with 95% confidence interval.
Time Frame: Up to 2 years
Population: Two patients were not evaluable for response due to rapid clinical deterioration
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 19
percentage of participants | 21 [6 to 46]

2. Secondary Outcome: Disease Control Rate
Description: Disease control rate is defined as N (%) patients with CR, PR, or SD by 24 weeks on study using RECIST version 1.1. For SD determination for DCR, the patient must have lack of progression for the first 24 weeks on study. Disease control rate will be assessed in the Response-evaluable and As-treated populations. Will be evaluated by RECIST version 1.1. Will be estimated with 95% confidence interval.
Time Frame: Up to 2 years
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
percentage of participants | 37 [16 to 62]

3. Secondary Outcome: Median Progression Free Survival (PFS)
Description: Progression Free Surival is defined as time in months from start of study treatment to first documentation of objective tumor progression as assessed by RECIST v1.1; Will be summarized using the method of Kaplan and Meier and Cox proportional hazards models.
Time Frame: Up to 2 years
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
Months | 4.6 [2.8 to 7.2]

4. Secondary Outcome: Median Overall Survival
Description: Will be summarized using the method of Kaplan and Meier and Cox proportional hazards models.
Time Frame: Up to 2 years
Population: The cervical cancer cohort had 12 participants. The non cervical cohort had 9 participants.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Group
Number analyzed (Participants) | 21
months
  Entire Population | 17.7 [7.6 to NA] — upper limit of the confidence interval was not estimable due to an insufficient number of participants with events
  Cervical Cancer Cohort: number analyzed (Participants) | 12
  Cervical Cancer Cohort | 7.6 [3.7 to 17.7]
  Non Cervical Cohort: number analyzed (Participants) | 9
  Non Cervical Cohort | 0 [NA to NA] — insufficient number of participants with events

ADVERSE EVENTS:
Time Frame: From the first dose through 30 days after the last dose of study medication, up to 2 years
Arm/Group | Treatment Group
All-Cause Mortality (participants affected / at risk) | 2/21
Serious Adverse Events (participants affected / at risk) | 1/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=21)
Lipase increased (Investigations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=21)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase - increased (Investigations) | 5
Alkaline phosphatase - increased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Aspartate aminotransferase - increased (Investigations) | 4
Blood bilirubin increased (Investigations) | 2
CPK increased (Investigations) | 2
Cholecystitis (Hepatobiliary disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Creatinine increased (Investigations) | 1
Dizziness (Nervous system disorders) | 1
Dry mouth (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Eosinophilia (Investigations) | 1
Fatigue (General disorders) | 10
Fever (General disorders) | 1
Headache (Nervous system disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperthyroidism (Endocrine disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypothyroidism (Endocrine disorders) | 4
Injection site reaction (General disorders) | 20
Lipase increased (Investigations) | 4
Lymphopenia (Blood and lymphatic system disorders) | 3
Mucositis oral (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 1
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3
Serum amylase increased (Investigations) | 3
Sinus bradycardia (Cardiac disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/85/NCT03439085/Prot_SAP_000.pdf